CLINICAL TRIAL: NCT01113112
Title: Biobehavioral-Cytokine Interactions in Ovarian Cancer
Acronym: VEGF
Status: Completed | Type: Observational
Sponsor: Susan Lutgendorf (Other)
Collaborators: University of Iowa (Other); National Cancer Institute (NCI) (NIH); Washington University School of Medicine (Other)
Responsible Party: Sponsor-Investigator, Susan Lutgendorf, Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 200308061; R01CA104825 (NIH)
Record Dates: First submitted 2010-04-27; First posted 2010-04-29 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Ovarian Neoplasms
Keywords: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, saliva, tissue, ascites
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Biobehavioral factors: Those with biobehavioral factors that contribute to a permissive local environment for macrophage-tumor interactions that enhance tumor growth in ovarian cancer

SUMMARY:
The purpose of this study is to understand relationships between behavioral factors, hormones, and chemicals produced by the body that may help tumor growth in ovarian cancer.

DETAILED DESCRIPTION:
Ovarian cancer is the second most common gynecologic cancer. Because of low rates of survival for the majority of ovarian cancer patients, identification of factors contributing to tumor progression is of paramount importance. Epidemiologic studies have suggested an association between biobehavioral factors such as life stress, depression, low social support and cancer progression. Direct links have been demonstrated between biobehavioral factors and cytokines supporting angiogenesis, the formation of new blood vessels that enhance tumor growth and progression. However, little is known regarding tumor associated macrophages (TAM) and interactions between TAM tumor cells in a way that favors tumor growth, but there is preliminary data indicating that ovarian cancer patients with higher levels of depressive symptoms and life stress have greater TAM production of matrix metalloproteinase-9, a key molecule promoting angiogenesis and tumor invasion. We also have preliminary data that ovarian cancer patients with high levels of depressive symptoms accompanied by low social support have greater tumor expression of a number of genes related to inflammation and tumor progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologic diagnosis of epithelial ovarian cancer, primary peritoneal carcinoma, or fallopian tube cancer; FIGO stage I to IV defined surgically at the completion of the initial abdominal surgery and with appropriate tissue available for histologic evaluation.
* Patients with the following histologic epithelial cell types are eligible: serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell carcinoma, mixed epithelial carcinoma, or adenocarcinoma not otherwise specified. However, the histologic features must be compatible with primary Mullerian epithelial adenocarcinoma.
* GOG performance status 0-3

Exclusion Criteria:

* Patients with a diagnosis of borderline epithelial ovarian tumor (formerly: tumors of low malignant potential" or recurrent invasive epithelial ovarian, primary peritoneal, or fallopian tube cancer treated with chemotherapy or radiotherapy previously are excluded.
* Patients who received neoadjuvant chemotherapy for ovarian, primary peritoneal, or fallopian tube carcinoma are excluded.
* Non-epithelial ovarian cancers or metastases to the ovaries from organs are excluded.
* Previous cancer diagnosis except for basal cell carcinoma of the skin or history of lymphoma.
* Pregnancy or age <18 years old
* Use of systemic glucocorticoids such as prednisone or decadron in the last 30 days
* Comorbid conditions: Addison's disease, autoimmune hepatitis, hepatitis B, hepatitis C, AIDS or HIV, lupus erythematosus, mixed connective tissue disease, rheumatoid arthritis.
* Inability to accurately answer questions (e.g. a condition such as dementia)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gyn/Onc patients at the University of Iowa and Washington University School of Medicine
Sampling Method: Non-Probability Sample
Enrollment: 613 (Actual)
Dates: Start 2003-08 (Actual); Primary Completion 2015-11-10 (Actual); Study Completion 2026-01-02 (Actual)

PRIMARY OUTCOMES:
Biobehavioral Factors | 1 year post op
  Pathways by which biobehavioral factors contribute to a permissive local environment for macrophage-tumor interactions that enhance tumor growth in ovarian cancer

CONTACTS AND LOCATIONS:
Overall Officials: Susan Lutgendorf, Ph.D., Principal Investigator — University of Iowa; Premal Thaker, MD, Study Chair — Washington University School of Medicine
Locations (2):
- United States (2):
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No